CLINICAL TRIAL: NCT03120104
Title: Physical Exercise for Colorectal Cancer Patients After Transanal Total Mesorectal Excision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201610007
Record Dates: First submitted 2017-04-05; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention group (Active Comparator): Pre-intervention group interventions:pelvic floor muscle training for one month (2~3 times a week, for 4 weeks) just one month before the stoma closure
  Interventions: Other: pelvic floor muscle exercise before stoma closure
- Post-intervention group (Active Comparator): Post-intervention group: pelvic floor muscle training for one month (2~3 times a week, for 4 weeks) two weeks after the stoma closure
  Interventions: Other: pelvic floor muscle exercise after stoma closure

INTERVENTIONS:
Other: pelvic floor muscle exercise before stoma closure — pelvic floor muscle training for one month (2~3 times a week, for 4 weeks) just one month before the stoma closure
  Arms: Pre-intervention group
Other: pelvic floor muscle exercise after stoma closure — pelvic floor muscle training for one month (2~3 times a week, for 4 weeks) just two weeks after the stoma closure
  Arms: Post-intervention group

SUMMARY:
Fecal incontinence is common in patients with rectal cancer after surgery. Previous studies showed that pelvic floor muscle and external sphincter muscle training after stoma closure could improve the severity of incontinence and other fecal symptoms, but there is no study about the effects of pelvic floor muscle exercise intervention before stoma closure. We are wondering would the symptom of fecal incontinence recover sooner and better if we give the pelvic floor muscle exercise intervention before the stoma closure. This article aims at comparing the effects of pelvic floor muscle training before stoma closure on fecal incontinence (pre-intervention group) with pelvic floor muscle training after stoma closure (post-intervention group), and we hypothesise that the severity of fecal incontinence will improve sooner and better in pre-intervention group.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer patients who have received transanal total mesorectal excision(TaTME) surgery; 20~75 years old

Exclusion Criteria:

* terminal stage of cancer; unable to following orders due to poor cognitive condition; too weak to follow the experimental procedures; central nervous system lesions

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change of The Wexner Score | measurement point 1: 2 weeks after the stoma closure; measurement point 2: 1 month after the intervention start
  for the change of severity of fecal incontinence assessment

SECONDARY OUTCOMES:
Change of St. Mark's Hospital Incontinence Score | measurement point 1: 2 weeks after the stoma closure; measurement point 2: 1 month after the intervention start
  for the change of severity of fecal incontinence assessment
Change of Functional assessment of Cancer Therapy - Colorectal (FACT-C) | measurement point 1: 2 weeks after the stoma closure; measurement point 2: 1 month after the intervention start
  for the change of quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Pin Li, Principal Investigator — Rehabilitation Department of Taipei Municipal WanFang Hospitial (Managed by Taipei Medical University)
Locations (1):
- Taipei Municipal Wanfang Hospital (Managed by Taipei Medical University), Taipei, Taiwan